CLINICAL TRIAL: NCT05013099
Title: A Phase IIB, Open Label, Study of Zirconium Zr 89 Crefmirlimab Berdoxam PET/CT in Subjects With Advanced or Metastatic Malignancies, Scheduled to Receive Immunotherapy (IOT) as a Single Agent or Combination, to Predict Response to Therapy
Brief Title: Study of Zirconium Zr 89 Crefmirlimab Berdoxam PET/CT in Subjects With Advanced or Metastatic Malignancies
Acronym: iPREDICT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IAB-CD8-203
Record Dates: First submitted 2021-07-30; First posted 2021-08-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Melanoma; Merkel Cell Carcinoma, Unspecified; Renal Cell Carcinoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with melanoma, Merkel cell, renal cell, or NSCLC (Experimental): Eligible subjects will receive up to three zirconium Zr 89 crefmirlimab berdoxam PET scans (up to 1.0 mCi ± 20% at 1.5 mg API per scan, for a total of up to 3.0 mCi ± 20% and 4.5 mg API) as an IV infusion or slow bolus injection as follows: First scan within 14 days prior to the onset of IOT, and a second scan 4 to 6 weeks after start of immunotherapy. The second zirconium Zr 89 crefmirlimab berdoxam administration and scan should be completed prior to the start of the third cycle of IOT. Subjects who are determined by the treating physician to have PD on immunotherapy can receive the optional third zirconium Zr 89 crefmirlimab berdoxam PET scan at the principal investigator's (PI's) discretion.
  Interventions: Biological: zirconium Zr 89 crefmirlimab berdoxam

INTERVENTIONS:
Biological: zirconium Zr 89 crefmirlimab berdoxam — Up to three zirconium Zr 89 crefmirlimab berdoxam PET scans (up to 1.0 mCi ± 20% at 1.5 mg API per scan, for a total of up to 3.0 mCi ± 20% and 4.5 mg API) as an IV infusion or slow bolus injection as follows: First (PETbaseline) within 14 days prior to the onset of IOT, and a second (PETEOC1) 4 to 6 weeks after start of immunotherapy. The second zirconium Zr 89 crefmirlimab berdoxam administration and scan (PETEOC1) should be completed prior to the start of the third cycle of IOT. Subjects who are determined by the treating physician to have PD on immunotherapy can receive the optional third zirconium Zr 89 crefmirlimab berdoxam PET scan at the principal investigator's (PI's) discretion.
  Other Names: 89Zr-Df-crefmirlimab; 89Zr-Df-IAB22M2C

SUMMARY:
The purpose of this study is to evaluate whether zirconium Zr 89 crefmirlimab berdoxam (other names 89Zr-crefmirlimab berdoxam, 89Zr-Df-crefmirlimab, 89Zr-Df-IAB22M2C) PET/CT can predict the response of advanced or metastatic melanoma, Merkel cell carcinoma, renal cell carcinoma, or non-small cell lung cancer tumors to immuno-oncology therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for enrollment in the study if they meet ONE criteria a, b or c in point 1 and ALL the criteria in points 2-9.

  1. Subjects must meet ONE of the criteria a, b or c below:

     1. For enrollment into Cohort A: Subjects with histologically confirmed advanced or metastatic non-uveal/non-mucosal melanoma or merkel cell carcinoma (MCPyV positive and negative) who are not amenable to surgical cure and are candidates to receive single- or combined IOT alone (not to include cytotoxic chemotherapy) as first or second line treatment.
     2. For enrollment into Cohort B: Subjects with histologically confirmed advanced or metastatic clear cell Renal Cell Carcinoma or Renal Cell Carcinoma with sarcomatoid features (regardless of subtype) as defined on pathologic examination by a component of clear cell or sarcomatoid, who are not amenable to surgical cure and are candidates to receive single- or combined IOT alone or IOT in combination with VEGFR-directed or tyrosine kinase inhibitor (not to include cytotoxic chemotherapy) as first or second line treatment
     3. For enrollment into Cohort C: Subjects with histologically confirmed advanced or metastatic non-small cell lung cancer without non-smoker/driver mutations who are not amenable to surgical cure, and are candidates to receive single- or combined IOT alone (not to include cytotoxic chemotherapy) as first or second line treatment as per the label/prescribing information at the physicians discretion.

     i. Patients with driver mutations that are expected to show significant benefit from first line checkpoint inhibiter treatment (such as KRAS G12C mutations) are eligible if all other I/E criteria are met

     Subjects must meet All of the criteria 2-9 below:
  2. At least 1 RECIST 1.1-measurable. non-irradiated, non-osseous (unless there is an associated measurable soft-tissue component) lesion documented on intravenous (IV) contrast-enhanced CT or MRI (per RECIST criteria 1.1) prior to first zirconium Zr 89 crefmirlimab berdoxam administration.
  3. Has an adequate amount of time between their prior treatment/procedure and the 1st administration of zirconium Zr 89 crefmirlimab berdoxam.
  4. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 and anticipated survival of at least 6 months.
  5. Meeting all clinical safety lab values per institution's SOC, or investigator's discretion, for subjects receiving cancer treatment.
  6. Male or female age ≥18 years.
  7. Ability to understand the purposes and risks of the trial and has signed an Institutional Review Board (IRB) approved informed consent form.
  8. Willingness and ability to comply with all protocol required procedures.
  9. For men and women of child-producing potential, use of effective double barrier contraceptive methods during the study, up to 30 days after the last administration of the investigational product.

Exclusion Criteria:

* Subjects will NOT be eligible for enrollment in the study if they meet ANY of the following criteria:

  1. Bone-only disease without a measurable soft tissue component on conventional imaging (MRI, PET, CT).
  2. Subjects with skin-only (cutaneous) lesions will be excluded from the tumor biopsy assessment.
  3. Serious nonmalignant disease, additional active malignant disease or conditions that in the opinion of the investigator and/or ImaginAb could compromise protocol objectives.
  4. Subjects with splenic dysfunction or who are status post splenectomy. Post-splenectomy subjects who develop an accessory spleen with clinical and radiographic evidence of splenic function will be allowed with prior approval from the Sponsor.
  5. Corticosteroid therapy is prohibited if used for the treatment of inflammatory or autoimmune conditions. Patients with adrenal insufficiency from prior surgery or immunotherapy toxicity may be on standard chronic replacement doses of hydrocortisone that also require sporadic use of stress doses of steroid .
  6. Pregnant women or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Best overall response (BOR) assessed by conventional imaging CT and/or MRI using RECIST 1.1 tomography/computed tomography (PET/CT) | Baseline to at least 24 or 27 weeks after the start of IOT, depending on treatment schedule.
  Best overall response (BOR) assessed by conventional imaging CT and/or MRI using RECIST 1.1 from 3 (or up to 3) consecutive imaging assessments (CT and/or MRI) following onset of immuno-oncology treatment.

SECONDARY OUTCOMES:
Largest measured difference from baseline in the lesion major axis from three (or up to three) consecutive standard of care imaging assessments (CT and/or MRI) | Baseline to at least 24 or 27 weeks after the start IOT, depending on treatment schedule.
  Largest measured difference from baseline in the lesion major axis from three (or up to three) consecutive standard of care imaging assessments (CT and/or MRI) following onset of immuno-oncology treatment.
Incidence and severity of AEs | Up to 48 weeks or end of treatment.
  Incidence and severity of AEs
Incidence and severity of infusion or injection reactions | 33 days post infusion
  Incidence and severity of infusion or injection reactions reported during or shortly after administration of the investigational product.
Incidence of withdrawal from scanning protocol due to zirconium Zr 89 crefmirlimab berdoxam related AEs | Up to 48 weeks or end of treatment
  Incidence of withdrawal from scanning protocol due to zirconium Zr 89 crefmirlimab berdoxam related AEs
12-lead ECG ventricular rate (bpm) | baseline to 48 weeks or end of study
  Ventricular rate (bpm) will be recorded from the 12-lead ECG
12-lead ECG PR interval (msec) | baseline to 48 weeks or end of study
  PR interval (msec) will be recorded from the 12-lead ECG
12-lead ECG QRS interval (msec) | baseline to 48 weeks or end of study
  QRS interval (msec) will be recorded from the 12-lead ECG
12-lead ECG QT interval (msec) | baseline to 48 weeks or end of study
  QT interval (msec) will be recorded from the 12-lead ECG
12-lead ECG QTc interval (msec) | baseline to 48 weeks or end of study
  QTc interval (msec) will be recorded from the 12-lead ECG
12-lead ECG Overall Result | baseline to 48 weeks or end of study
  Investigator's overall assessment of the ECG reading will be recorded as normal or abnormal. If abnormal, as either "not clinically significant" or "clinically significant"
Anti-drug antibody | baseline to 48 weeks or end of study
  Detection of anti-drug antibodies
Change in blood AST levels (U/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood AST levels (U/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood ALT levels (U/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood ALT levels (U/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood ALP levels (U/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood ALP levels (U/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood bilirubin levels (mg/dL) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood bilirubin levels (mg/dL) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood LDH levels (U/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood LDH levels (U/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood BUN levels (mg/dL) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood BUN levels (mg/dL) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood GGT levels (U/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood GGT levels (U/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in serum creatinine levels (mg/dL) from baseline. | Baseline through 48 weeks or end of treatment.
  Serum creatinine levels (mg/dL) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood uric acid levels (mg/dL) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood uric acid levels (mg/dL) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood sodium levels (mmol/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood sodium (mmol/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood potassium levels (mmol/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood potassium (mmol/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood chloride levels (mmol/L) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood chloride (mmol/L) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.
Change in blood glucose levels (mg/dL) from baseline. | Baseline through 48 weeks or end of treatment.
  Blood glucose (mg/dL) will be obtained at baseline and collected prior to each administration and 60 minutes post administration.

OTHER OUTCOMES:
Evaluate zirconium Zr 89 crefmirlimab berdoxam PET/CT as a discriminator of pseudo-progression. | Up to 48 weeks or end of treatment.
  Incidence of iRECIST defined pseudo-progression events.
Evaluate zirconium Zr 89 crefmirlimab berdoxam PET/CT in subjects who develop clinical and/or radiographic progression to explore mechanisms for treatment resistance. | Up to 48 weeks or end of treatment.
  RECIST 1.1 defined Progressive Disease.
Evaluate zirconium Zr 89 crefmirlimab berdoxam PET/CT as a predictor or surrogate for IOT immune related adverse events (irAEs). | Up to 48 weeks or end of treatment.
  Incidence of Immuno-oncology related TEAEs in non-diseased tissues and organs.
Correlate zirconium Zr 89 crefmirlimab berdoxam PET uptake with CD8 expression and PD 1/PD-L1 expression as determined by immunohistochemistry (IHC). | Up to 48 weeks or end of treatment.
  CD8 expressing cells and PD-1/PD-L1 expressing cells.
Evaluate zirconium Zr 89 crefmirlimab berdoxam PET/CT as a predictor of progression free survival (PFS) | Up to 48 weeks or end of treatment.
  Patient level Progression Free Survival.
Evaluate zirconium Zr 89 crefmirlimab berdoxam PET/CT as a predictor of duration of response (DoR). | Up to 48 weeks or end of treatment.
  Patient level Duration of Response.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Margolin, MD, Principal Investigator — Providence Saint John's Cancer Institute
Locations (16):
- United States (6):
  - CARTI Cancer Center, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Providence Saint John's Cancer Institute, Santa Monica, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- Australia (5):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Olivia Newton-John Cancer Research Insititute, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- University Hospitals Leuven, Leuven, Belgium
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Leiden University Medical Center, Leiden
- Lausanne University Hospital, Lausanne, Switzerland
- Northern Centre for Cancer Care and Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No